CLINICAL TRIAL: NCT03483857
Title: Peer Navigation to Improve Engagement in Care for HIV-Positive Men Who Have Sex With Men in Ehlanzeni, South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: ANOVA Health Institute (Unknown); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R34MH109395-01 (NIH)
Record Dates: First submitted 2017-10-24; First posted 2018-03-30 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Hiv
Keywords: Peer Navigation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Two arm study assessing to determine feasibility and acceptability of a pilot PN intervention among 100 HIV-positive MSM. We will explore associations between PN participation and continuum of care outcomes in a cohort of 55 HIV-positive MSM receiving PN, as compared to a cohort of 48 HIV-positive MSM receiving standard-of-care clinical referral, in preparation for a full-scale multi-site behavioral efficacy trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Navigation (Experimental): Individuals assigned to the PN condition will be assigned to one of 10 PN case managers who will follow an SOP described for initial intake and follow up visits with each participant. Participants will be asked to provide contact information for themselves and up to 3 individuals whom study staff can contact in case they cannot make direct contact with the study participant assigned to PN. PN will meet with their clients at least once monthly to discuss treatment related issues including medication access, side effects, adherence, stigma or discrimination related to HIV or their taking ART medication, etc. Participants will have contact information for their assigned PN and may contact them for reasons related to their treatment between scheduled monthly visits if they choose. All visits with PN will be recorded by the PN. and participants who fail to attend up to 3 scheduled PN appointments will be considered LTFU for the intervention.
  Interventions: Behavioral: Peer Navigation
- Standard of Care (No Intervention): Individuals assigned to SOC will be referred directly to the NCHC/RLS staff for treatment initiation or continuation. At intake they will receive standard treatment information per MPDOH guidelines, as well as information about Anova's RLS and Health4Men clinical and psychosocial services available at the NCHC. They will receive monthly text message reminders from study staff to refill ART prescriptions, and a separate reminder in month 6 to schedule complete their 6-month clinical visit. Study staff will verify that participants have picked up medications and attended all scheduled clinical visits by means of chart review and data extraction. Per MPDOH guidelines, individuals who fail to collect medications 3 months in a row, or who fail to attend their 6-month HIV clinical follow-up appointment, will be considered non-engaged and lost to follow up (LTFU).

INTERVENTIONS:
Behavioral: Peer Navigation — Utilizing Peer Navigators for HIV-Positive MSM for increase in uptake along the continuum.
  Arms: Peer Navigation

SUMMARY:
This protocol describes the Cohort Assessment phase of an R34 pilot intervention trial of a Peer Navigation (PN) intervention tailored to the needs of HIV-positive MSM in rural Mpumalanga province South Africa. The PN intervention to be adapted, I-Care, has been implemented among HIV-positive men and women in the general population in North West province, South Africa, by members of this research team.

ELIGIBILITY:
Inclusion Criteria:

* Biological male;
* Age >=18 years;
* Self-identify as a gay or bisexual man, or a transgender woman;
* Have male sexual partners within the prior six months
* Resident in the Ehlanzeni District Municipality for at least six months of the year;
* Be physically present in Ehlanzeni for at least two weeks per month
* Self-disclosed receiving an HIV-positive diagnosis in the last 5 years;
* Consent to all serological testing for HIV antibodies, ART analytes, and HIV RNA
* Consent for study staff to review participants' clinical records;
* Consent to the randomization process.

Exclusion Criteria:

* Inability to provide written informed consent for participation, including being under the influence of alcohol or drugs.
* Inability to provide laboratory or documentary evidence of HIV diagnosis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — As this study focuses on men who have sex with men, only persons born male are included.
Enrollment: 103 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
Viral Suppression | 6 months
  The proportion of participants virally suppressed (HIV RNA <1000 copies/microliter) in Peer Navigation (Intervention) arm compared to standard of care (SOC) arm.

CONTACTS AND LOCATIONS:
Overall Officials: Sheri Lippman, PhD, Principal Investigator — University of California, San Francsico
Locations (1):
- Anova Health Institute, Mbombela, Mpumalanga, South Africa

IPD SHARING:
Plan to Share IPD: No